CLINICAL TRIAL: NCT02873897
Title: Acceptability of Products and Eating Pleasure in Elderly People Living at Home or in an EHPAD
Brief Title: Acceptability of Products and Eating Pleasure in Elderly People Living at Home or in Establishment Hosting For the Dependant Elderly (EHPAD) (Old-people's Home)
Acronym: OPTIFEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: VAN WYMELBEKE FP7 2012
Record Dates: First submitted 2016-08-04; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Nutrition
Keywords: elderly

ARMS (2):
- Group "meals on wheels at home" (Other)
  Interventions: Dietary Supplement: Experimental session: to select enriched products; Dietary Supplement: Control session
- Group "residents of old people's homes - EHPAD (Other)
  Interventions: Dietary Supplement: Session A: Experimental products (selected enriched products); Dietary Supplement: Session B: Control (standard products without enrichment)

INTERVENTIONS:
Dietary Supplement: Session A: Experimental products (selected enriched products)
  Arms: Group "residents of old people's homes - EHPAD
Dietary Supplement: Experimental session: to select enriched products
  Arms: Group "meals on wheels at home"
Dietary Supplement: Session B: Control (standard products without enrichment)
  Arms: Group "residents of old people's homes - EHPAD
Dietary Supplement: Control session
  Arms: Group "meals on wheels at home"

SUMMARY:
In independent elderly people, the aim is to test recipes for different types of food from different countries (starter, main course with culinary aids, carrot purees, desserts and smoothies) likely to improve sensory acceptability of foods for elderly people who are dependent for their meals (persons for whom at least one meal per day is provided by a catering service - meals at home, old people's home). All of the recipes were developed thanks to the first two parts of the OPTIFEL project so as to take into account the needs of elderly people and recommendations in each country. The interest is to increase the sapidity/ attractiveness of meals by optimizing sensory properties and the nutritional content of the foods, to meet the nutritional needs of this specific population with enriched recipes (with leguminous proteins and/or vitamins and minerals and/or fibre) suitable for different cultures. This ongoing research is being conducted on 2-4 different variants of each type of product: the starter (a soup of legumes), the main dish (diced chicken with culinary aids) and garnished (carrot puree), an apple-based dessert and fruit smoothies.

For each product family, two products will be selected for each country: the preferred product (highest hedonic value of recipes enriched with leguminous proteins and/or vitamins and minerals) and the standard product without enrichment.

Finally, at the end of this study, nine products will have been chosen: 2 soups, 2 culinary aids, 2 carrot purees, 2 desserts and 1 smoothie

ELIGIBILITY:
Inclusion Criteria:

* people older than 65 years
* persons living in EHPAD-type old people's homes or living at home and using a meals-on-wheels service
* persons without known heart disease or arterial hypertension
* persons who have given oral consent

Exclusion Criteria:

* Persons suffering from a serious illness during the trial
* Persons with life expectancy of less than 6 months
* Persons with proven anosmia (total loss of olfaction), from birth or because of physical trauma (head injury) or disease (acute rhinitis)
* Persons with an allergy or an aversion for any of the foods used
* Persons with a strict prescribed diet

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Measuring new product satisfaction | throughout the study; completion up to 13 months
  Measure satisfaction with new products developed and chosen for elderly people living at home with meals-on wheels or in EHPAD (old people's homes)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France